CLINICAL TRIAL: NCT06115590
Title: Novel Objective Digital Biomarkers for Assessing Sub-clinical Mood Disturbances in the Singaporean Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Human Development and Potential (IHDP), Singapore (Other)
Collaborators: OBVIO HEALTH USA, Inc. (Unknown)
Responsible Party: Principal Investigator, Jeroen Schmitt, Senior Principal Investigator, Institute for Human Development and Potential (IHDP), Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-018
Record Dates: First submitted 2023-10-23; First posted 2023-11-03 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Mood
Keywords: Digital Biomarkers; Mood; Stress; Mental Health
MeSH Terms: conditions — Psychological Well-Being | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: 8-day parallel-group design with decentralized data collection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Stress (No Intervention): Reference Group
- Elevated Stress (No Intervention): Half of the Participants(n=40) with elevated stress (PSS score >13) will be randomly assigned to this group
- Elevated Stress intervention (Experimental): Half of the Participants(n=40) with High stress (PSS score >13) will be randomly assigned to this group
  Interventions: Dietary Supplement: Nutritional supplement

INTERVENTIONS:
Dietary Supplement: Nutritional supplement — Nutritional intervention hypothesized to have an acute anxiolytic effect
  Arms: Elevated Stress intervention

SUMMARY:
The investigators aim to assess the relationship between objectives markers (of physiological reactivity) recorded using a smartwatch and self-reported subjective outcomes measured using standardized and non-standardized questionnaires recorded in an eDiary; with stress as the model for our assessment utilizing the validated PSS-10 questionnaire.

As personal characteristics such as personality traits, resilience, and grit have been shown to modulate reactivity and mental health status, the investigators aim to explore the modulation of the study outcomes by such personality factors. Furthermore, the investigators aim to explore the association of the study outcomes with the composition and functional potential of the gut microbiome.

Finally, the investigators aim to explore the effects of a nutritional intervention on our outcome measures.

Participants will participate in a decentralized, parallel-group study with a mixed design lasting 8 days (excluding screening and enrollment). A total of 120 participants are divided into low-stress(n=40), and elevated-stress groups (n=80) based on their perceived stress score (PSS-10, cut-off score 13). A subgroup of elevated-stress participants (n=40) will be administered a nutritional intervention for 3 days. Their responses will be compared to another subgroup of elevated-stress participants (n=40) without intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 to 30 years
* Own and uses a smartphone that is capable of running the study applications
* Have access to the internet
* Adequate fluency in the English language to understand the informed consent process, study instructions and study assessments
* Sufficient vision and hearing to complete study procedures
* Willing to commit to about 20 minutes of assessments each day for a period of 8 days
* Willing to wear selected study devices 24 hours/day; 7-days per week with only occasional relief
* Willing and able to participate and to give written informed consent

Exclusion Criteria:

* Past (< 6 months prior to the study) or current neurological or psychiatric condition
* Past (< 3 months prior to the study) or current use of psychoactive medication
* Having received antibiotic treatment < 4 weeks prior to the study
* Present or past history of alcohol or drug addiction and/or recreational drug use
* Maltodextrin allergy
* Members of the research team or their immediate family members. An immediate family member is defined as spouse, parent, child, or sibling, whether biological or legally adopted
* Women participants who are currently pregnant or have been pregnant in past 6 months

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2024-02-18 (Actual); Study Completion 2024-02-18 (Actual)

PRIMARY OUTCOMES:
Depression Anxiety and Stress Scale 21 (DASS-21) | 7 days
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self- report scales designed to measure the emotional states of depression, anxiety and stress in clinical and non-clinical populations. Each of the three DASS-21 scales contains 7 items that are scored on a 4-point Likert scale (0-3). In the current study a modified version is used where subjects rate their symptoms over the past 24 hours, rather than 1 week.
  This questionnaire will be completed daily at 9 pm.
State Trait Anxiety Inventory (STAI-6) 23 | 7 days
  The STAI-6 is a validated short-form version (6 items) of the 40-item STAI questionnaire, measuring current anxiety symptoms on a 4-point Likert scale. Total score is calculated (range 6-24).
  This questionnaire will be completed daily at 1 pm.

SECONDARY OUTCOMES:
Ecological Momentary Assessment | 7 days
  In the smartphone application, subject will be prompted four times a day with the following statements. The EMA assessment will occur daily at 9.00 am, 1.00 pm, 5.00 pm, 9.00 pm. Subjects are asked to indicate their current state on a VAS (Visual analog Scale). The score in the scale ranges from 0 to 100. 0 being "Not at all" and 100 being "Very Much".
  The participants will be asked to respond to the following questions:
  "Right now, I feel mentally sharp" - to assess perception of cognitive ability "Right now, I feel fatigued" - to assess fatigue/exhaustion directly "Right now, I feel stressed" - to assess stress "Right now, I feel nervous" - to assess nervousness/tension "Right now, I feel depressed" - to assess depression "Right now, I am in a good mood" - to assess joy "Right now, I feel thirsty" - to assess level of thirst "Right now, I feel hungry" - to assess level of hunger "I slept well last night" - to assess subjective sleep quality
Activity | 7 days
  Activity level, including #steps, distance traveled, and floors climbed, is measured using a Fitbit Sense 2 smart watch.
Respiratory rate | 7 days
  Respiratory rate (breaths per minute) is measured using a Fitbit Sense 2 smart watch.
Heart rate | 7 days
  Heart rate (beats per minute) is continuously measured using a Fitbit Sense 2 smart watch.
Sleep | 7 days
  Sleep duration (minutes) and quality are measured using a Fitbit Sense 2 smart watch.
Blood oxygenation level (SpO2) | 7 days
  Blood oxygenation level (%) is measured using a Fitbit Sense 2 smart watch.
Electrodermal activity (EDA) | 7 days
  In four user-initiated 2-min sessions per day, Electrodermal activity is measured via a Fitbit Sense 2 smart watch.

OTHER OUTCOMES:
Stool microbiome composition | baseline
  Stool samples will be collected at home on the first test day and analyzed for gut microbiome composition using shotgun metagenomic sequencing.
stool microbiome functional potential | baseline
  In addition to mapping the taxonomic abundance, the gut microbiome functional potential will be analysed using Biobakery analysis tools.

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore Institute for Clinical Trials, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No